CLINICAL TRIAL: NCT00583414
Title: Endovascular Exclusion of Abdominal Aortic Aneurysms in High Risk Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Federico Ezequiel Parodi, Staff, The Cleveland Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G980198; IRB 3264 (Other: Cleveland Clinic IRB)
Record Dates: First submitted 2007-12-20; First posted 2007-12-31 (Estimated); Results first posted 2019-01-25 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Abdominal Aortic Aneurysm; Iliac Aneurysm; Internal Iliac Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Iliac Aneurysm | interventions — Endovascular Aneurysm Repair

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Endovascular Aneurysm Repair (Experimental): Investigational stent-graft implant to exclude aneurysm
  Interventions: Device: Endovascular Aneurysm Repair

INTERVENTIONS:
Device: Endovascular Aneurysm Repair — Endovascular exclusion of aneurysm
  Other Names: Cook Zenith

SUMMARY:
The purpose of this study is to assess the role of abdominal aneurysm and iliac aneurysm exclusion using an endovascular prosthesis.

DETAILED DESCRIPTION:
This study is a prospective, non-randomized evaluation of endovascular aneurysm repair in high-risk patients. The purpose of this study is to determine whether this endovascular prosthesis is safe and effective for the intended use of treating AAA/iliac aneurysm in patients who are at high risk for standard aneurysm surgical repair. Up to 400 patients will be enrolled at the Cleveland clinic Foundation. Baseline procedures may include angiogram, intravascular ultrasound, CT scan, physical exam, blood work and ankle-brachial index. The endovascular prosthesis is placed in the operating room under regional or general anesthesia and the procedure length is approximately 2-3 hours. Follow up evaluations will be done at 1 month, 6 months (if clinically necessary), 12 months and yearly, and may include a physical exam, CT scan, KUB, ultrasound, blood work, and an ankle-brachial index.

ELIGIBILITY:
Inclusion Criteria:

* The aneurysm is >/= 5 cm or larger, or with a high risk of rupture due to its shape, history of growth, symptoms, or the presence of a large (>2 cm) iliac aneurysm
* Anticipated mortality greater than 10 percent with conventional surgery
* Life expectancy greater than 2 years
* Suitable arterial anatomy
* Absence of systemic disease or allergy that precludes an endovascular repair
* Capable of giving informed consent and willingness to comply with the follow-up schedule

Exclusion Criteria:

* Pregnancy
* History of anaphylactic reaction to contrast material with an inability to properly prophylax the patient appropriately
* Allergy to stainless steel or polyester
* Unwilling to comply with the follow-up schedule
* Serious or systemic groin infection
* Coagulopathy, other than coumadin therapy
* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 401 (Actual)
Dates: Start 1998-09 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Eagleton, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Farivar BS, Abbasi MN, Dias AP, Kuramochi Y, Brier CS, Parodi FE, Eagleton MJ. Durability of iliac artery preservation associated with endovascular repair of infrarenal aortoiliac aneurysms. J Vasc Surg. 2017 Oct;66(4):1028-1036.e18. doi: 10.1016/j.jvs.2017.02.042. Epub 2017 May 11. PMID 28502545
- [Derived] Eagleton MJ, Shah S, Petkosevek D, Mastracci TM, Greenberg RK. Hypogastric and subclavian artery patency affects onset and recovery of spinal cord ischemia associated with aortic endografting. J Vasc Surg. 2014 Jan;59(1):89-94. doi: 10.1016/j.jvs.2013.07.007. Epub 2013 Nov 1. PMID 24188715

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Endovascular Aneurysm Repair
Started | 401
Completed | 401
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Endovascular Aneurysm Repair
Number analyzed (Participants) | 401
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 56
  >=65 years | 345
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 358
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Presence of AAA or Iliac Aneurysm [Number; unit: participants] | 401

OUTCOME MEASURES:

1. Primary Outcome: Freedom From Aneurysm Rupture
Description: Absence of blood extravasation outside of aneurysm sac demonstrated by CT scan
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Endovascular Aneurysm Repair
Number analyzed (Participants) | 401
Participants | 0

ADVERSE EVENTS:
Time Frame: At discharge, 1-, 6-, 12- and 24-month.
Arm/Group | Endovascular Aneurysm Repair
All-Cause Mortality (participants affected / at risk) | 292/401
Serious Adverse Events (participants affected / at risk) | 9/401
Other Adverse Events (participants affected / at risk) | 9/401
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Endovascular Aneurysm Repair (N=401)
Aneurysm Growth (Vascular disorders) | 9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Endovascular Aneurysm Repair (N=401)
Aneurysm Growth (Vascular disorders) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2002-10-04): https://cdn.clinicaltrials.gov/large-docs/14/NCT00583414/Prot_SAP_ICF_000.pdf